CLINICAL TRIAL: NCT03622853
Title: What Factors Area Associated With Prognosis After Steroid Hydrodilatation for Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02-005c
Record Dates: First submitted 2018-03-29; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis
MeSH Terms: conditions — Bursitis | interventions — Steroids

STUDY DESIGN:
Intervention Model Description: To investigate the factors associated with improvement after intraarticular steroid injection for patients with Frozen shoulder
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intraarticular steroid injection (Experimental): intraarticular steroid hydrodilatation (shincort 40mg )
  Interventions: Drug: Steroid (shincort)

INTERVENTIONS:
Drug: Steroid (shincort) — intraarticular shincort 40mg / 4ml mixed with 2% xylocaine and Normal saline
  Other Names: shincort

SUMMARY:
To investigate the factors associated with improvement after intraarticular steroid injection for patients with Frozen shoulder

DETAILED DESCRIPTION:
Objective: To investigate the factors associated with improvement after intraarticular steroid injection for patients with Frozen shoulder

Design: Prospective study.

Participants: Patients with Frozen shoulder were recorded the demographic data, associated disease, ultrasound findings at baselines.

Intervention: One shot intraarticular steroid hydrodilatation

Main Outcome Measures: Visual analog scale (VAS) of the shoulder pain, Constant score, SPADI score, and angles of active and passive shoulder range of motion (flexion, abduction, external rotation, and internal rotation) at pre-treatment, post-treatment at week 8

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of frozen shoulder by physical examination and ultrasonography

Exclusion Criteria:

1. other conditions involving the shoulder ( rheumatoid arthritis, Hill-Sachs lesions,osteoporosis, or malignancies in the shoulder region);
2. neurologic deficits affecting shoulder function in normal daily activities;
3. shoulder pain caused by cervical radiculopathy
4. a history of drug allergy to xylocaine
5. pregnancy or lactation;
6. received injection into the affected shoulder during the preceding 3 months

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
The change of constant shoulder score between week 0 and week 8 | 0 and 8 wks
  the total constant score ranges from 0 to 100 points, with higher scores indicative of better function. The score is divided into four sections: pain, activity of daily living, ROM and strength

SECONDARY OUTCOMES:
pain intensity | 0 and 8 wks
  pain intensity was measured by visual analog scale. Each patient was asked to indicate his/her current level of pain by marking a point on a 100-mm VAS, for which 0 represented no pain and 100 represented unbearable pain.
Shoulder Pain And disability index | 0 and 8 wks
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
glenohumeral joint range of motion | 0 and 8 wks
  Shoulder flexion, abduction, external rotation and internal rotation were measured with goniometer with patient in supine position

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No